CLINICAL TRIAL: NCT03930212
Title: Progesterone Supplementation in Threatened Abortion: Is it a Sound Practice?
Brief Title: Progesterone Supplementation in Threatened Abortion
Acronym: Prothreat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Prog133077
Record Dates: First submitted 2019-04-20; First posted 2019-04-29 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Threatened Abortion; Progesterone Resistance
MeSH Terms: conditions — Abortion, Threatened; Progesterone Resistance | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progesterone (Experimental): received rectal progesterone suppositories 400 mg once daily
  Interventions: Drug: Progesterone
- Control group (Placebo Comparator): received placebo suppositories rectally once daily.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Progesterone — received rectal progesterone suppositories 400 mg once daily
  Arms: Progesterone
Drug: Placebos — received placebo suppositories rectally once daily.
  Arms: Control group

SUMMARY:
To decide whether progesterone supplementation in threatened abortion is a sound practice.

DETAILED DESCRIPTION:
This study was conducted at Obstetrics and Gynecology Department, Tanta University in the period from January 2018 to December 2018. Patients: Eligible patients (n=190) were randomly allocated into 2 groups; study group who will receive progesterone supplementation (Prog.group) and control group who will receive no treatment (place.group).

ELIGIBILITY:
Inclusion Criteria:

* threatened abortion diagnosed by history and ultrasound examination
* singleton
* viable fetus
* gestational age < 20 weeks
* closed normal length cervix.

Exclusion Criteria:

* short cervix <2 cm Multiple pregnancy
* dead fetus
* open cervix ≥ 2cm
* history of cervical surgery
* refusal to participate.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
relief of pain | 3 weeks
  questionnaire fulfilled by patient with yes or no questions
completion of pregnancy beyond 20 weeks | 12 weeks
  passing the age 20 weeks
Stoppage of bleeding | 3 weeks
  Cessation of bleeding

SECONDARY OUTCOMES:
abortion less than 20 weeks. | 12 weeks
  Abortion

CONTACTS AND LOCATIONS:
Locations (1):
- Ayman Shehata Dawood, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 2 months